CLINICAL TRIAL: NCT03469323
Title: Can Mini-dose Succinylcholine Accelerate Lung Collapse and Intrathoracic Nerve Blocks During Nonintubated Thoracoscopic Surgery? A Randomized Controlled Trial
Brief Title: Effects of Succinylcholine on Nonintubated Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 201711080MINB
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Tumor of Lung Parenchyma; Complication of Ventilation Therapy; Atelectasis
Keywords: Nonintubated video-assisted thoracic surgery (VATS)
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Succinylcholine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonintubated VATS succinylcholine (Experimental): Nonintubated VATS using mini-dose succinylcholine in the beginning of open pneumothorax
  Interventions: Drug: Succinylcholine
- Nonintubated VATS placebo (Placebo Comparator): Nonintubated VATS not using succinylcholine in the beginning of open pneumothorax
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Succinylcholine — Giving mini-dose succinylcholine to facilitate lung collapse during nonintubated VATS.
  Other Names: Suxamethonium
  Arms: Nonintubated VATS succinylcholine
Drug: Placebo — Giving placebo (normal saline) to facilitate lung collapse during nonintubated VATS.
  Other Names: Normal saline
  Arms: Nonintubated VATS placebo

SUMMARY:
A safe and effective surgical environment is important for nonintubated thoracoscopic surgery. The investigators hypothesize that mini-dose succinylcholine can induce ultra-short period of apnea, by which the ventilatory responses to open pneumothorax were abolished and may facilitate rapid and satisfying collapse of the operated lung during nonintubated thoracoscopic surgery.

DETAILED DESCRIPTION:
Background: Nonintubated thoracoscopic surgery is the frontier of modern minimal invasive thoracic surgery. A safe and effective surgical environment is established via an iatrogenic open pneumothorax producing the operated lung fully collapsed. However, the initial respiratory response to open pneumothorax is both tachypnea and carbon dioxide rebreathing, which would jeopardize the quality of collapse of the operated lung and delay the performance of intrathoracic vagal block. Intravenous opioid is effective to attenuate ventilatory responses but herein with risk of persistent respiratory depression.

Methods: The investigators hypothesize that mini-dose succinylcholine 0.15 mg/kg can induce ultra-short period of apnea, by which the ventilatory responses to open pneumothorax were abolished and may facilitate rapid and satisfying collapse of the operated lung during nonintubated thoracoscopic surgery. In a prospective, randomized, double-blind study design, 30 patients will be allocated to receive either succinylcholine (n=15) or placebo (n=15) in the beginning of open pneumothorax. The effectiveness of succinylcholine will be measured by the surgeon's evaluation of the quality of lung collapse, while the safety will be evaluated by determination of arterial blood gases within 20 minutes of one-lung spontaneous breathing.

Expected results: Mini-dose succinylcholine can facilitate early lung collapse without jeopardizing the ventilatory function during nonintubated thoracoscopic surgery with one-lung spontaneous breathing, which may make nonintubated thoracoscopic surgery easier and safer.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with lung tumors and elective for unilateral thoracoscopic surgery.

Exclusion Criteria:

* Over weighted, body mass index > 26 kg/m2.
* Previous thoracic surgery on the attempted operative side.
* Hypoventilation syndrome requiring positive pressure ventilatory support or oxygen at home.
* Relevant systemic disease, including heart failure, liver failure, renal failure with an American Society of Anesthesiologists (ASA) class above 3.
* Difficult airway management.
* Pregnancy.
* Contraindications for succinylcholine, including family history of suspicious malignant hyperthermia, hyperkalemia, or other neuromuscular diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of lung collapse | 20 minutes
  Quality of lung collapse will be quantified by the surgeon as score 1-3.

SECONDARY OUTCOMES:
Arterial blood gas analysis | 20 minutes
  Arterial partial pressure of carbon dioxide (PaCO2) and oxgen (PaO2) levels after succinylcholine and placebo during one-lung ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hui Hung, MD, MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan